CLINICAL TRIAL: NCT01845974
Title: Atrial Pressure Electrophysiology Pilot Study: Comparison of High vs. Low Flow Catheters During Radiofrequency Catheter Ablation (RFCA) for Atrial Fibrillation (AF).
Brief Title: Atrial Pressure Electrophysiology Pilot Study
Acronym: APES
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim evaluation of data after internal safety report from sponsor.
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: #5387
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2018-01

CONDITIONS: Atrial Fibrillation
Keywords: Radiofrequency Catheter Ablation; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Flow Catheter (Experimental): The experimental group will receive the low flow catheter (ThermoCool® SF NAV Catheter) All data will be collected pre and post procedure therefore patients will act as their own control within each therapeutic group.
  Interventions: Device: ThermoCool® SF NAV Catheter
- High Flow Catheter (Active Comparator): The control group will receive the higher flow catheter (ThermoCool® catheter). All data will be collected pre and post procedure therefore patients will act as their own control within each therapeutic group.
  Interventions: Device: ThermoCool® catheter

INTERVENTIONS:
Device: ThermoCool® SF NAV Catheter — The experimental group will receive the low flow catheter (ThermoCool® SF NAV Catheter) All data will be collected pre and post procedure therefore patients will act as their own control within each therapeutic group.
  Arms: Low Flow Catheter
Device: ThermoCool® catheter — The control group will receive the higher flow catheter (ThermoCool® catheter). All data will be collected pre and post procedure therefore patients will act as their own control within each therapeutic group.
  Arms: High Flow Catheter

SUMMARY:
This study examined data elements of hemodynamic, electrophysiologic and electrolyte trends comparing 2 different types of catheters used during a procedure to treat medication resistant atrial fibrillation-radiofrequency catheter ablation. A high flow catheter delivers a high volume of saline during the procedure. The low flow catheter delivers a low volume of saline during the procedure. The patient will be consented and randomized to one of the 2 groups using a computer generated randomization chart. Those that are put in the low flow catheter group will be considered the experimental group. All data will be collected before and after the procedure and each patient will act as their own control within each group.

DETAILED DESCRIPTION:
Final report

ELIGIBILITY:
Inclusion Criteria:

* Drug resistant paroxysmal AF
* ≥ 18 years old

Exclusion Criteria:

* Left atrial thrombus on TEE
* Patients unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Miller, MD, Principal Investigator — Advocate Lutheran General Hospital
Locations (1):
- Advocate Lutheran General Hospital, Park Ridge, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kiraly LN, Differding JA, Enomoto TM, Sawai RS, Muller PJ, Diggs B, Tieu BH, Englehart MS, Underwood S, Wiesberg TT, Schreiber MA. Resuscitation with normal saline (NS) vs. lactated ringers (LR) modulates hypercoagulability and leads to increased blood loss in an uncontrolled hemorrhagic shock swine model. J Trauma. 2006 Jul;61(1):57-64; discussion 64-5. doi: 10.1097/01.ta.0000220373.29743.69. PMID 16832250
- [Background] Antoniou A, Milonas D, Kanakakis J, Rokas S, Sideris DA. Contraction-excitation feedback in human atrial fibrillation. Clin Cardiol. 1997 May;20(5):473-6. doi: 10.1002/clc.4960200514. PMID 9134280
- [Background] Ninio DM, Saint DA. Passive pericardial constraint protects against stretch-induced vulnerability to atrial fibrillation in rabbits. Am J Physiol Heart Circ Physiol. 2006 Nov;291(5):H2547-9. doi: 10.1152/ajpheart.01248.2005. Epub 2006 Jun 23. PMID 16798819
- [Background] Satoh T, Zipes DP. Unequal atrial stretch in dogs increases dispersion of refractoriness conducive to developing atrial fibrillation. J Cardiovasc Electrophysiol. 1996 Sep;7(9):833-42. doi: 10.1111/j.1540-8167.1996.tb00596.x. PMID 8884512
- [Background] Gupta A, Lawrence AT, Krishnan K, Kavinsky CJ, Trohman RG. Current concepts in the mechanisms and management of drug-induced QT prolongation and torsade de pointes. Am Heart J. 2007 Jun;153(6):891-9. doi: 10.1016/j.ahj.2007.01.040. PMID 17540188

RESULTS

PARTICIPANT FLOW:
Recruitment Details: all patients scheduled for atrial fibrillation ablation referred to study coordinator. Non qualifying reasons include: Clot on TEE;Persistant AFib despite previous treatments;Combo treatment needed for both atrial fibrillation and flutter; Declined participation:Afib the morning of procedure;ICD;Rhythm other than Sinus Rhythm
Period: Overall Study
Arm/Group | Low Flow Catheter | High Flow Catheter
Started | 4 | 9
Completed | 3 | 9
Not Completed | 1 | 0
Not completed — screen failure | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Flow Catheter | High Flow Catheter | Total
Number analyzed (Participants) | 4 | 9 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (16.5) | 61.3 (9) | 61.23 (11.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 2 | 6 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 9 | 13
Comorbidities [Count of Participants; unit: Participants]
  Hypertension | 2 | 5 | 7
  Heart Failure | 2 | 0 | 2
  Diabetes | 1 | 2 | 3
  Obstructive sleep apnea | 3 | 1 | 4
  Coronary artery disease | 2 | 2 | 4
Tobacco history [Count of Participants; unit: Participants] | 0 | 5 | 5
Previous therapies [Count of Participants; unit: Participants]
  statin | 2 | 4 | 6
  angiotensin 2 receptor blockers | 1 | 2 | 3
  angiotensin converting enzymes | 0 | 3 | 3
  beta blockers | 2 | 7 | 9
  digoxin | 0 | 2 | 2
  spiranolactone | 0 | 0 | 0
  diuretic | 1 | 0 | 1
CHADsVasc 2 score= 2+ [Count of Participants; unit: Participants] — Congestive heart failure = 1 Hypertension: blood pressure consistently above 140/90 mmHg (or treated hypertension on medication) =1; Age ≥75 years=2 Diabetes Mellitus =1; Prior Stroke or TIA or thromboembolism =2 ;Vascular disease (e.g. peripheral artery disease, myocardial infarction, aortic plaque) =1; Age 65-74 years =1; Sex category female =+1-items are summed to arrive at a score ranging from 0 to 9, with scores >=2 indicating "moderate-high" stroke risk".)
  Participants | 3 | 9 | 12
prior cardiac surgery [Count of Participants; unit: Participants]
  pacemaker | 0 | 1 | 1
  coronary artery bypass grafting | 0 | 1 | 1
  surgical maze | 0 | 0 | 0
  right atrial flutter ablation | 0 | 2 | 2
  prior catheter Radiofrequency ablation for Afib | 1 | 2 | 3
Prior Antiarrhythmia drug failure [Count of Participants; unit: Participants]
  none | 0 | 1 | 1
  sotolol | 1 | 1 | 2
  dofetilide | 0 | 1 | 1
  fleccainide | 0 | 2 | 2
  dronedarone | 1 | 3 | 4
  ammiodarone and fleccainide | 1 | 0 | 1
  ammiodarone and dronedarone | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hemodynamic, Electrolyte, and Electrophysiologic Derangements
Description: The objective of this pilot study is to investigate the use of a lower flow catheter (ThermoCool® SF NAV Catheter, Biosense Webster, Inc. Diamond Bar, CA, eluting 8-15ml/minute during RF lesion delivery) vs. a higher flow catheter (ThermoCool® catheter, same manufacturer, eluting 17-30 ml/minute), Outcomes are measured by number of Participants with Hemodynamic, Electrolyte, and Electrophysiologic Derangements, is reported. This was measured as participants requiring electrolyte replacement, if the BP dropped below 100 mm in CICU or if participants sustained atrial tachyarrhythmias
Time Frame: Observation period is up to the 24 hours post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Low Flow Catheter | High Flow Catheter
Number analyzed (Participants) | 3 | 9
Participants
  Required electrolyte replacement | 2 | 6
  patients withSystolic BP < 100 mm in CIC | 1 | 5
  sustained atrial tachyarrhythmias | 0 | 1

ADVERSE EVENTS:
Time Frame: 24 hours post procedure
Arm/Group | Low Flow Catheter | High Flow Catheter
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/9
Other Adverse Events (participants affected / at risk) | 0/4 | 0/9

LIMITATIONS AND CAVEATS:
early termination due to safety memo issued by sponsor

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other